CLINICAL TRIAL: NCT05072821
Title: Immediate Injection of Botulinum Toxin Type a After Keloid Scar Revision to Prevent Keloid Recurrence: a Prospective, Split-scar, Double-blind, Randomized Controlled Study
Brief Title: Botulinum Toxin Type a Injection to Prevent Keloid Recurrence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Tainan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MOHW109-TDU-B-211-114003
Record Dates: First submitted 2021-08-30; First posted 2021-10-11 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Scar Keloid
Keywords: Keloid; Botulinum Toxin type A; Radiotherapy
MeSH Terms: conditions — Keloid | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum Toxin type A injection side (Experimental): The Botulinum Toxin type A will be injected into the dermal layer before skin closure in keloid excision surgery. The concentration of Botulinum Toxin type A is 100 units in 2 mL and dosage is 8 units/cm. The maximal dose is 100 units for each participant.
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]
- 0.9% saline injection side (Placebo Comparator): The 0.9% saline will be injected into the dermal layer before skin closure in keloid excision surgery. The dosage is 0.16 mL/cm.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [Botox] — After the whole surgical procedures of keloid revision are done, the participants will receive Botulinum Toxin type A (BTA) injection. The investigators split the scar into the right side and the left side. BTA and 0.9% saline, respectively, are used for the two arms of the study. Vials containing 100 units of BTA (BotoxⓇ, Allergan) are mixed with 2mL 0.9% injectable saline. The injection depth will be the intradermal layer. Injections will be performed with a 30-gauge needle and 1 mL syringe. Just before skin closure, the entire scar was treated, with sides randomized to receive treatment with either BTA or 0.9% normal saline. The dosage is 8 units / cm based on aforementioned studies. The maximal dose won't exceed 100 units.
  Arms: Botulinum Toxin type A injection side
Drug: 0.9% Sodium Chloride Injection — After the whole surgical procedures of keloid revision are done, the participants will receive 0.9% saline injection. The investigators split the scar into the right side and the left side. BTA and 0.9% saline, respectively, are used for the two arms of the study. Only 0.9% saline is injected on the control side. The injection depth will be the intradermal layer. Injections will be performed with a 30-gauge needle and 1 mL syringe. Just before skin closure, the entire scar was injected, with sides randomized to receive treatment with either BTA or 0.9% normal saline. The dosage is 0.16 mL / cm.
  Arms: 0.9% saline injection side

SUMMARY:
The prospective, split-scar, double-blind, randomized controlled study will enroll the patients who are older than 20 years with progressive keloid lesion which is symmetric. Botulinum toxin A will be injected into half of each keloid revision wound immediately after skin closure. The scars will be assessed at 1-year follow-up with Vancouver Scar Scale (VSS), Patient and Observer Scar Assessment Scale (POSAS), and the Cutometer.

DETAILED DESCRIPTION:
Continuous variables will be reported as the mean ± standard deviation(SD). Each aspect of the VSS score, POSAS score, and the Cutometer parameters of each scar half between the BTA and control groups will be analyzed longitudinally using the paired t test. The interrater consistency will be evaluated using the Spearman rho. All analyses will be performed with IBM SPSS Version 23.0 (IBM Corp., Redmond, Wash.). A value of p < 0.05 is considered to indicate statistical significance.

The sample size was calculated based on the results of the investigators' aforementioned study published in 2019. Thirty patients underwent keloid revision and then received radiation therapy based on our treatment protocol. The postoperative Vancouver Scar Scale score was 4.15 ± 1.74. If treatment could improve VSS score by 1, which was considered clinically significant, approximately 26 patients would have been necessary to provide a result with a real significance (using the same SD and considering the standard α error of 0.05 and a power of 0.8). Assuming a 20% non-compliance rate for follow-up evaluation, the sample size was increased to 32 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (20 years or older)
* Progressive keloid lesion that is bilaterally symmetric, mandibular area, anterior chest or suprapubic area, for example
* At least 4 cm in length
* Repeated or uncontrolled recurrence, and unendurable symptoms with poor response to conservative modalities
* Valid written informed consent provided for surgery and trial inclusion

Exclusion Criteria:

* Allergy to botulinum toxin
* Previous botulinum toxin injection at the lesion within 6 months before enrollment
* Myasthenia gravis
* Focal infection signs
* Pregnant or breastfeeding woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Keloid recurrence | One year
  The recurrence of keloid will be determined by clinical examination evaluated by a dermatologist.

SECONDARY OUTCOMES:
Subjective symptoms | 3, 6, 9 and 12 months
  The subjective symptoms will be measured by the Patient Scale of the Patient and Observer Scar Assessment Scale. The Patient Scale consists six items and scores from 1 to 10 for each items. The score of 1 means much alike the normal skin and the score of 10 means worst imaginable scar.
Objective symptoms | 3, 6, 9 and 12 months
  The subjective symptoms will be measured by the Observer Scale of the Patient and Observer Scar Assessment Scale. The Observer Scale consists six items and scores from 1 to 10 for each items. The score of 1 means much alike the normal skin and the score of 10 means worst imaginable scar.
Vancouver Scar Scale | 6 and 12 months
  One dermatologist will evaluate the scar with the Vancouver Scar Scale. The Vancouver Scar Scale consists 4 items. The minimum score is 0, which means the scar is much alike normal skin. The maximal score is 13, which means purple, hyperpigmentation, contracture and elevated scar.
Scar firmness | 6 and 12 months
  The scar firmness is determined by the Cutometer parameter R0. R0 is maximum amplitude of the curve (the total elongation). The larger R0 is, the softer the scar is.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Yu Hsueh, MD PhD, Principal Investigator — National Cheng-Kung University and Hospital
Locations (1):
- National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan, Taiwan